CLINICAL TRIAL: NCT05963113
Title: A Single-center Randomized Clinical Trial to Test the Efficacy of Pharyngeal Swallowing Exercises (With or Without Protein Supplementation) to Build Pharyngeal Muscular Reserve in Pre-frail Older Adults
Brief Title: Pharyngeal Exercise (Plus Protein)
Acronym: PE(PP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 23-00293
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Pre-Frail Older Adults
Keywords: proactive exercise; protein; nutrition

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI, outcome assessors, and individuals conducting data analyses will be blinded to randomization. The treating clinicians and participants will be aware of their study group given that they will be provided with either water or protein drinks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control, then Swallowing Exercises + Protein (Experimental): Participants randomized to 12 weeks of swallowing exercises with protein supplementation, after completing an initial 12-week period of "usual activity."
  Interventions: Behavioral: Pharyngeal Swallowing Exercises; Dietary Supplement: Protein Supplementation; Device: MRI
- Control, then Swallowing Exercises (Active Comparator): Participants randomized to 12 weeks of swallowing exercises without protein supplementation, after completing an initial 12-week period of "usual activity."
  Interventions: Behavioral: Pharyngeal Swallowing Exercises; Device: MRI

INTERVENTIONS:
Behavioral: Pharyngeal Swallowing Exercises — 12-weeks of proactive pharyngeal swallowing exercises conducted 5 times per week. The exercise program will include the following four exercises: effortful saliva swallows, tongue-hold swallows, effortful pitch glides and posterior lingual resistance. Each exercise set will include 10 repetitions of each exercise (40 reps per set). The number of sets will be gradually increased as tolerance builds.
Dietary Supplement: Protein Supplementation — 12-week supply of the commercially-available Premier Protein Clear ® High Protein (20 grams of protein and 90 calories per 16.9 oz. drink). Participants will be asked to consume one drink per day for the 12-week intervention period.
  Arms: Control, then Swallowing Exercises + Protein
Device: MRI — Participants will be scanned using a 3T MRI scanner and a 16-channel phased array neck coil.

SUMMARY:
The swallowing muscles are prone to decreased strength and function as part of the natural aging process which can lead to difficulty swallowing, malnutrition, and frailty. Exercise and nutrition are powerful stimulators of muscular change. The proposed research will investigate the effectiveness of a 12-week proactive regimen of swallowing exercises (with or without daily protein supplement drinks) to improve the composition, force, and physiology of the swallowing muscles and explore the relationship to overall health and physical function in 80 community-dwelling older adults. Each participant will serve as their own control for 12 weeks before being randomized to complete swallowing exercises alone or swallowing exercises with protein drinks.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 65 years of age or older.
2. Participants must score a 1 or 2 on the FRAIL scale OR a 4 or greater on the Strength, Assistance in Walking, Rise from a Chair, Climb Stairs and Falls (SARC-F) Questionnaire.
3. Participants must score 26 or greater on the Montreal Cognitive Assessment (MoCA).
4. Willingness to participate in the study procedures.

Exclusion Criteria:

1. Known structural or neurological causes of dysphagia.
2. Cannot consume high levels of protein (Chronic Kidney Disease Stage 3 or higher).
3. Contraindications to 3T whole body MRI scanners (e.g., pacemaker, cerebral aneurysm clip, cochlear implant, presence of shrapnel in strategic locations, metal in the eye, claustrophobia, or other problems).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Thickness of the Superior Pharyngeal Constrictor Muscle | Baseline, Week 13
  Axial T2-weighted images through the C1 level, hyoid bone and arytenoid cartilages will be used to measure the thickness of the superior pharyngeal constrictor muscle.
Change in Thickness of the Superior Pharyngeal Constrictor Muscle | Baseline, Week 28
  Axial T2-weighted images through the C1 level, hyoid bone and arytenoid cartilages will be used to measure the thickness of the superior pharyngeal constrictor muscle.
Change in Thickness of the Middle Pharyngeal Constrictor Muscle | Baseline, Week 13
  Axial T2-weighted images through the C1 level, hyoid bone and arytenoid cartilages will be used to measure the thickness of the middle pharyngeal constrictor muscle.
Change in Thickness of the Middle Pharyngeal Constrictor Muscle | Baseline, Week 28
  Axial T2-weighted images through the C1 level, hyoid bone and arytenoid cartilages will be used to measure the thickness of the middle pharyngeal constrictor muscle.
Change in Thickness of the Inferior Pharyngeal Constrictor Muscle | Baseline, Week 13
  Axial T2-weighted images through the C1 level, hyoid bone and arytenoid cartilages will be used to measure the thickness of the inferior pharyngeal constrictor muscle.
Change in Thickness of the Inferior Pharyngeal Constrictor Muscle | Baseline, Week 28
  Axial T2-weighted images through the C1 level, hyoid bone and arytenoid cartilages will be used to measure the thickness of the inferior pharyngeal constrictor muscle.
Change in Maximum Pharyngeal Constriction During Swallowing | Baseline, Week 13
  Maximum pharyngeal constriction area (normalized to spine length) will be captured at the height of the swallow on videofluoroscopy.
Change in Maximum Pharyngeal Constriction During Swallowing | Baseline, Week 28
  Maximum pharyngeal constriction area (normalized to spine length) will be captured at the height of the swallow on videofluoroscopy.

SECONDARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) Scores | Baseline, Week 13
  The SPPB comprises a gait speed test, a chair stand test, and three balance tests. The gait speed test score ranges from 0 (worst outcome) to 4 (best outcome); the chair stand test score ranges from 0 (worst outcome) to 4 (best outcome); the side-by-side stand test score ranges from 1 (best outcome) to 0 (worst outcome); the semi-tandem stand test score ranges from 1 (best outcome) to 0 (worst outcome); and the tandem stand test scores range from 2 (best outcome) to 0 (worst outcome).
  The total SPPB score is the sum of the test scores and ranges from 0-12, with lower scores indicating greater disability.
Change in Short Physical Performance Battery (SPPB) Scores | Baseline, Week 28
  The SPPB comprises a gait speed test, a chair stand test, and three balance tests. The gait speed test score ranges from 0 (worst outcome) to 4 (best outcome); the chair stand test score ranges from 0 (worst outcome) to 4 (best outcome); the side-by-side stand test score ranges from 1 (best outcome) to 0 (worst outcome); the semi-tandem stand test score ranges from 1 (best outcome) to 0 (worst outcome); and the tandem stand test scores range from 2 (best outcome) to 0 (worst outcome).
  The total SPPB score is the sum of the test scores and ranges from 0-12, with lower scores indicating greater disability.
Change in Fat-Free Muscle Index | Baseline, Week 13
  Fat-free muscle index measured via bioelectrical impedance analysis using the InBody 570 multi-frequency analyzer.
Change in Fat-Free Muscle Index | Baseline, Week 28
  Fat-free muscle index measured via bioelectrical impedance analysis using the InBody 570 multi-frequency analyzer.
Change in Pre-Albumin Levels | Baseline, Week 13
  Levels of pre-albumin, a marked of undernutrition, will be measured using patient blood samples.
Change in Pre-Albumin Levels | Baseline, Week 28
  Levels of pre-albumin, a marked of undernutrition, will be measured using patient blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Molfenter, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Steinhardt School of Education, New York, New York
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: smm16@nyu.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to smm16@nyu.edu. To gain access, data requestors will need to sign a data access agreement.